CLINICAL TRIAL: NCT04577573
Title: Cognitive-based Rehabilitation Platform of Hand Grasp After Spinal Cord Injury Using Virtual Reality and Instrumented Wearables
Brief Title: Cognitive-based Prosthetics to Improve Grasp and Reaching After SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Stevens Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: B3582-P
Record Dates: First submitted 2020-09-14; First posted 2020-10-08 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries; Hand Weakness
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: At each visit, prototype cognitive prosthetic devices will be tested under 3 conditions:
  No feedback, simple feedback, and enhanced feedback. Outcomes will include time taken for successful movements; and accuracy of movements.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- No cognitive feedback (Active Comparator): Perform task without cognitive feedback.
  Interventions: Device: Cognition glove; Device: Sensory brace
- Intermediate feedback. (Active Comparator): Perform task with intermediate feedback.
  Interventions: Device: Cognition glove; Device: Sensory brace
- Enhanced feedback (Experimental): Perform task with virtual reality and/or haptic feedback.
  Interventions: Device: Cognition glove; Device: Sensory brace

INTERVENTIONS:
Device: Cognition glove — The investigators have developed and tested a functional prototype of an instrumented glove to alert the user about secure grasp of objects. Onboard force and flex sensors provide inputs to a machine learning algorithm (artificial neural network, ANN) to estimate secure grasp based on previously collected training data. The glove enhances agency by alerting the user to secure grasp through sensory feedback modules (visual - LED, audio - beeper, tactile - vibrator).
Device: Sensory brace — A a size- and position-adjustable arm brace with weight-support capability and housing for vibration motors and EMG sensors. Position adjustment allows for physical therapists to find and recommend arm postures that are clinically relevant to
  each person. The participant can then isometrically push/resist against the brace to strengthen target muscles while performing VR reach-to-touch. The person will receive visual feedback from the virtual environment to train movement performance and vibrotactile feedback at tendons to subconsciously adjust their muscle activation patterns

SUMMARY:
Rehabilitation of functional movements after spinal cord injury (SCI) requires commitment and engagement to the processes of physical therapy. Outcomes may be improved by techniques that strengthen cognitive connections between users and physical therapy exercises.

The investigators will investigate combinations of virtual reality and innovative wearable technology to accelerate rehabilitation of hand grasp and reach. These devices use multi-sensory feedback to enhance the sense of agency, or feelings of control, and better train movements during physical rehabilitation exercises. The investigators will measure the effect of these devices on improving the speed, efficiency, and accuracy of performed movements in Veterans with SCI.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) at the cervical level impairs hand function severely compromises performance of activities of daily living. The physical rehabilitation process requires commitment by the participant to achieve meaningful gains in function. Rehabilitation approaches that are cognitively engaging can facilitate greater commitment to practice and improved movement learning.

The investigators propose to develop innovative platforms that utilize virtual reality (VR) and instrumented wearables that enhance cognitive factors during motor learning of hand grasp and reach after SCI. These factors include greater sense of agency, or perception of control, and multi-sensory feedback. Sense of agency is implicated with greater movement control, and various sensory feedback modalities (visual, audio, and haptic) are proven effective in movement training. However, these factors are not well considered in traditional physical therapy approaches.

The investigators have developed two novel cognitive-based platforms for rehabilitating grasp and reach function and propose to test each platform in Veterans with chronic SCI at the cervical level.

Aim 1 will investigate how the "cognition" glove may improve functional grasp. This glove includes force and flex sensors that provide inputs to a machine learning algorithm trained to predict when secure grasp is achieved. The glove alerts the user of secure grasp through onboard sensory modules providing visual (LED), audio (beeper), and tactile (vibrator) feedback. During training, feedback is provided at gradually shorter time-intervals to progressively induce agency based on the neuroscience principle of 'intentional binding'. This principle suggests that with greater agency, one perceives their action (i.e., secure grasp) is more coupled in time to a sensory consequence (i.e., glove feedback). The glove is user-ready, and now has compatibility with customized VR applications to provide enhanced sensory feedback through engaging and customized visual and sound alerts. The investigators hypothesize that enhanced feedback in VR will produce even greater improvements in grasp performance than onboard feedback alone.

Aim 2 will investigate how Veterans with SCI may learn greater arm muscle control during virtual reaching while using a "sensory" brace that provides isometric resistance to one arm to elicit electromyography (EMG) patterns that can drive a virtual arm. The person receives visual feedback from VR and muscle tendon haptic feedback from the brace during training. Tendon stimulation can elicit movement sensations that modulate muscle activation patterns. The VR feedback will provide conscious movement training cues while vibration feedback will subconsciously elicit more distinct EMG patterns based on cluster analysis. The investigators hypothesize that the promotion of distinct EMG patterns, achieved by maximizing inter-cluster distances, will improve performance of a reach-to-touch task.

Importantly, the concept of strengthening cognitive agency and learning of movement using wearable technology, multi-sensory feedback, and virtual reality during physical training will be applicable to all forms of neuromuscular impairment, including stroke and traumatic brain injury in addition to SCI.

ELIGIBILITY:
Inclusion Criteria:

* SCI occurred greater than 12 months ago
* SCI occurred between levels C1-T1
* Hand weakness: score of 2, 3, or 4 out of 5 on manual muscle testing of finger extension, finger flexion, or finger abduction in either hand

Exclusion Criteria:

* History of other serious brain or spinal cord injuries
* History of seizures
* Ventilator dependence; open tracheostomy
* Use of medications that significantly lower seizure threshold
* History of significant cognitive deficits
* Open skin lesions over the face, neck, shoulders, arms, or hands
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noam Y. Harel, MD PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be shared in electronic format pursuant to a VA-approved Data Use Agreement.
  This will include all outcomes data and deidentified demographics.
  Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 CFR Part 1.466.
Supporting Information: Study Protocol
Time Frame: Upon publication.
Access Criteria: Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 CFR Part 1.466.

REFERENCES:
- [Result] Liu M, Wilder S, Sanford S, Saleh S, Harel NY, Nataraj R. Training with Agency-Inspired Feedback from an Instrumented Glove to Improve Functional Grasp Performance. Sensors (Basel). 2021 Feb 7;21(4):1173. doi: 10.3390/s21041173. PMID 33562342

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognition Glove: Participants wear an instrumented glove on one hand while performing reaching and grasping tasks.
- Sensory Brace: Participants wear an instrumented brace on one shoulder/upper arm while performing reaching and grasping tasks.
- Participated in Both Cognition Glove and Sensory Brace: Participated in both Cognition Glove and Sensory Brace experiments
Period: Overall Study
Arm/Group | Cognition Glove | Sensory Brace | Participated in Both Cognition Glove and Sensory Brace
Started | 4 | 7 | 2
No Feedback | 4 | 7 | 2
Glove Feedback | 4 | 0 | 2
Glove + Virtual Reality (VR) Feedback | 4 | 0 | 2
Brace + Visual Feedback | 0 | 7 | 0
Brace + Visual + Haptic Feedback | 0 | 7 | 0
Completed | 4 | 5 | 2
Not Completed | 0 | 2 | 0
Not completed — Technical - invalid protocol | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognition Glove | Sensory Brace | Participated in Both Cognition Glove and Sensory Brace | Total
Number analyzed (Participants) | 4 | 7 | 2 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 2 | 13
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 2 | 6 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 7 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1
  White | 4 | 5 | 2 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Time to Achieve Secure Grasp (Cognition Glove Only)
Description: Percent change in time (seconds) to achieve secure grasp. Lower time is better.
Time Frame: Baseline and Following the 6 hour lab session, assessed while performing the task
Population: Data invalid for one participant in No cognitive feedback, 2 participants in Intermediate feedback, and 1 participant in Enhanced feedback
Measure: Mean (Standard Deviation); unit: % change in time to secure grasp
Groups:
- No Cognitive Feedback: Perform task without cognitive feedback.
  Cognition glove: The investigators have developed and tested a functional prototype of an instrumented glove to alert the user about secure grasp of objects. Onboard force and flex sensors provide inputs to a machine learning algorithm (artificial neural network, ANN) to estimate secure grasp based on previously collected training data. The glove enhances agency by alerting the user to secure grasp through sensory feedback modules (visual - LED, audio - beeper, tactile - vibrator).
  Sensory brace: A a size- and position-adjustable arm brace with weight-support capability and housing for vibration motors and EMG sensors. Position adjustment allows for physical therapists to find and recommend arm postures that are clinically relevant to
  each person. The participant can then isometrically push/resist against the brace to strengthen target muscles while performing VR reach-to-touch. The person will receive visual feedback from the virtual environment to train movement performance and vibrotactile feedback at tendons to subconsciously adjust their muscle activation patterns
- Intermediate Feedback.: Perform task with intermediate feedback.
  Cognition glove: The investigators have developed and tested a functional prototype of an instrumented glove to alert the user about secure grasp of objects. Onboard force and flex sensors provide inputs to a machine learning algorithm (artificial neural network, ANN) to estimate secure grasp based on previously collected training data. The glove enhances agency by alerting the user to secure grasp through sensory feedback modules (visual - LED, audio - beeper, tactile - vibrator).
  Sensory brace: A a size- and position-adjustable arm brace with weight-support capability and housing for vibration motors and EMG sensors. Position adjustment allows for physical therapists to find and recommend arm postures that are clinically relevant to
  each person. The participant can then isometrically push/resist against the brace to strengthen target muscles while performing VR reach-to-touch. The person will receive visual feedback from the virtual environment to train movement performance and vibrotactile feedback at tendons to subconsciously adjust their muscle activation patterns
- Enhanced Feedback: Perform task with virtual reality and/or haptic feedback.
  Cognition glove: The investigators have developed and tested a functional prototype of an instrumented glove to alert the user about secure grasp of objects. Onboard force and flex sensors provide inputs to a machine learning algorithm (artificial neural network, ANN) to estimate secure grasp based on previously collected training data. The glove enhances agency by alerting the user to secure grasp through sensory feedback modules (visual - LED, audio - beeper, tactile - vibrator).
  Sensory brace: A a size- and position-adjustable arm brace with weight-support capability and housing for vibration motors and EMG sensors. Position adjustment allows for physical therapists to find and recommend arm postures that are clinically relevant to
  each person. The participant can then isometrically push/resist against the brace to strengthen target muscles while performing VR reach-to-touch. The person will receive visual feedback from the virtual environment to train movement performance and vibrotactile feedback at tendons to subconsciously adjust their muscle activation patterns
Arm/Group | No Cognitive Feedback | Intermediate Feedback. | Enhanced Feedback
Number analyzed (Participants) | 5 | 4 | 5
% change in time to secure grasp | 39.9 (65.5) | -14.6 (11.9) | 10.1 (54.9)

2. Primary Outcome: Percent Change in Time to Complete Pick-up and Placement of Object-Cognition Glove
Description: Percent change in time (seconds) to pick up and re-place object. Lower time is better.
Time Frame: Baseline and Following the 6 hour lab session, assessed while performing the task
Measure: Mean (Standard Deviation); unit: % change in time to pick-up/placement
Groups:
- Cognition Glove-No Feedback: Participants wear an instrumented glove on one hand while performing reaching and grasping tasks. No augmented feedback provided.
- Cognition Glove-Glove Feedback: Participants wear an instrumented glove on one hand while performing reaching and grasping tasks. Augmented feedback from the glove provided.
- Cognition Glove-VR Feedback: Participants wear an instrumented glove on one hand while performing reaching and grasping tasks. Augmented feedback from the glove and from virtual reality provided.
Arm/Group | Cognition Glove-No Feedback | Cognition Glove-Glove Feedback | Cognition Glove-VR Feedback
Number analyzed (Participants) | 6 | 6 | 6
% change in time to pick-up/placement | 20.2 (19.7) | 7.9 (25.8) | -24.4 (24.3)

3. Primary Outcome: Percent Change in Time to Complete Trial-Sensory Brace
Description: Percent change in time (seconds) to complete target reaching trials in VR environment. Lower time is better.
Time Frame: Baseline and Following the 6 hour lab session, assessed while performing the task
Population: Data invalid for two participants in each condition.
Measure: Mean (Standard Deviation); unit: % change in time to complete trial
Groups:
- Sensory Brace-Visual VR Feedback: Participants wear an instrumented brace on one shoulder/upper arm while performing reaching and grasping tasks. Augmented visual VR feedback from the brace provided.
- Sensory Brace-Haptic Plus Visual VR Feedback: Participants wear an instrumented brace on one shoulder/upper arm while performing reaching and grasping tasks. Augmented haptic plus visual VR feedback from the brace provided.
Arm/Group | Sensory Brace-Visual VR Feedback | Sensory Brace-Haptic Plus Visual VR Feedback
Number analyzed (Participants) | 5 | 5
% change in time to complete trial | 18.6 (9.1) | 3.3 (12.5)

4. Secondary Outcome: Percent Change in Motion Pathlength in Moving Object-Cognition Glove
Description: Percent change in pathlength during reaching/grasping/moving. Shorter is better.
Time Frame: Baseline and Following the 6 hour lab session, assessed while performing the task
Measure: Mean (Standard Deviation); unit: % change in motion pathlength
Arm/Group | Cognition Glove-No Feedback | Cognition Glove-Glove Feedback | Cognition Glove-VR Feedback
Number analyzed (Participants) | 6 | 6 | 6
% change in motion pathlength | 39.1 (13.1) | 21.9 (31.2) | -12.4 (19.1)

5. Secondary Outcome: Percent Change in Motion Pathlength Toward Virtual Targets-Sensory Brace
Description: Percent change in pathlength during reaching virtual targets. Shorter is better.
Time Frame: Baseline and Following the 6 hour lab session, assessed while performing the task
Population: Data invalid for two participants in each condition.
Measure: Mean (Standard Deviation); unit: % change in motion pathlength
Arm/Group | Sensory Brace-Visual VR Feedback | Sensory Brace-Haptic Plus Visual VR Feedback
Number analyzed (Participants) | 5 | 5
% change in motion pathlength | 17.7 (10.6) | 1.4 (6.5)

6. Secondary Outcome: Error in Placing Object Onto Target (Cognition Glove Only)
Description: Error in completing placement of object onto target.
Time Frame: Baseline and Following the 6 hour lab session, assessed while performing the task
Population: After initiating the study, it was quickly determined that this outcome measure was irrelevant. All participants are able to complete the task. Outcome measures 1 and 2 capture the impact of difficulty grasping and moving the object without requiring a separate subjective measure of 'error'.
Measure: Mean (Standard Deviation); unit: Error in placing object onto target.
Arm/Group | Cognition Glove-No Feedback | Cognition Glove-Glove Feedback | Cognition Glove-VR Feedback
Number analyzed (Participants) | 6 | 6 | 6
Error in placing object onto target. | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 24 hours.
Description: Participants were asked a standardized set of questions to review potential symptoms and adverse events.
Groups:
- Cognition Glove: Participants wear an instrumented glove on one hand while performing reaching and grasping tasks.
  Note, the 3 different feedback conditions all occur during the same session and involve wearing the same sensors, so it's not possible to distinguish condition-specific AEs, especially because no AEs occurred in this group.
- Sensory Brace: Participants wear an instrumented brace on one shoulder/upper arm while performing reaching and grasping tasks.
  Note, the 2 different brace feedback conditions all occur during the same session and involve wearing the same sensors, so it's not possible to distinguish the EEG cap-related discomfort according to feedback condition.
Arm/Group | Cognition Glove | Sensory Brace
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognition Glove (N=6) | Sensory Brace (N=7)
Discomfort from EEG gel in hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of participants in this pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT04577573/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT04577573/ICF_000.pdf